CLINICAL TRIAL: NCT04199039
Title: The Effects of Endotracheal Tube Fixation Methods on Hemodynamic Parameters During Endotracheal Suction in Cardiovascular Surgery Intensive Care Patients
Brief Title: Effects of Endotracheal Tube Fixation Methods on Hemodynamic Parameters During Endotracheal Suction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulay ALTUN UGRAS, Associate Professor, Mersin University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gulay altun ugras
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Cardiac Surgery
Keywords: endotracheal tube; nursing

STUDY DESIGN:
Intervention Model Description: prospective, single-blind non-randomized clinical trial study
Who Masked: Participant
Masking Description: In this study only the patient was blinded. Investigators involved with the running of the study were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET fixation with ET holder (Experimental): ET fixation of the patients in the study group was performed with an ET holder when they arrived at the CVS ICU
  Interventions: Other: Effect on Endotracheal Tube Fixation Methods on Hemodynamic Parameters During Endotracheal Suction
- ET fixation with plaster (No Intervention): ET fixation in the control group was performed with plasters, which are routinely used in the ICU where the study was conducted.

INTERVENTIONS:
Other: Effect on Endotracheal Tube Fixation Methods on Hemodynamic Parameters During Endotracheal Suction — When the study started, the first 43 patients were assigned to the control group and the following 43 patients were assigned to the study group in the CVS ICU. ET fixation in the control group was performed with plasters, which are routinely used in the ICU where the study was conducted. ET fixation of the patients in the study group was performed with an ET holder (AnchorFast Oral Endotracheal Tube Fastener, Hollister, Liberlyville, USA) when they arrived at the CVS ICU.
  The patients' SBP, DBP, HR and SpO2 values, which were displayed on the bedside monitor (Nihon Kohden, Tokyo), were recorded on the "Hemodynamic Parameters Form" just before, during, and at the end of endotracheal suction, and in the following 5th and 15th minutes.
  Arms: ET fixation with ET holder

SUMMARY:
Background: Endotracheal suction (ES), may cause changes like increase in blood pressure, heart rate (HR) and decrease in peripheral oxygen saturation (SpO2), which may cause changes in hemodynamic parameters (HPs) that increase the workload of the heart after surgery.

Aim: The aim of this study is to determine the effect of the methods used in endotracheal tube (ET) fixation on HPs [systolic blood pressure (SBP), diastolic blood pressure (DBP), HR and SpO2] during ES.

Study Design: The sample of this prospective, single-blind non-randomized clinical trial study included 86 intubated patients who were treated in the cardiovascular surgery intensive care unit (CVSICU) of a university hospital between September 2016 and December 2017.

Methods: The ET fixations of the experimental group (n=43) were performed with tube holders while the ET fixations of the control group (n=43) were performed using plasters. The HPs of the patients were measured before, during, at the end of suction and 5 and 15 minutes after suction.

DETAILED DESCRIPTION:
Information collected from the relatives of the patient, patient file and the health care workers was used to fill out the "Patient Information Form".

When the study started, the first 43 patients were assigned to the control group and the following 43 patients were assigned to the study group in the CVS ICU. ET fixation in the control group was performed with plasters, which are routinely used in the ICU where the study was conducted. ET fixation of the patients in the study group was performed with an ET holder (AnchorFast Oral Endotracheal Tube Fastener, Hollister, Liberlyville, USA) when they arrived at the CVS ICU.

When the findings of patients' suction needs were observed (increase in respiratory rate, HR increase, arterial BP increase, high pressure alarm in ventilator, mucus in ET, cyanosis, dyspnea, restlessness, sweating, disturbance of blood gas parameters, wheezing, etc.), endotracheal suction was performed according to the application standards. The patients' SBP, DBP, HR and SpO2 values, which were displayed on the bedside monitor (Nihon Kohden, Tokyo), were recorded on the "Hemodynamic Parameters Form" just before, during, and at the end of endotracheal suction, and in the following 5th and 15th minutes.

During the suction process, it was ensured that the patients were in the supine position in which the head of the bed was lifted by 30 degree Before the intra-arterial BP was measured, the transducer was reset at the level of the right atrial (plebostatic axis) and the position was not changed during all the measurements.

ELIGIBILITY:
Inclusion Criteria:

* postcardiac surgery
* having endotracheal tube

Exclusion Criteria:

- pulmonary problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | During the suction process
  systolic blood pressure (SBP), diastolic blood pressure (DBP), mmHg
Heart rate | During the suction process
  beats per minute
peripheral oxygen saturation | During the suction process
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

IPD SHARING:
Plan to Share IPD: No